CLINICAL TRIAL: NCT06426667
Title: Effect of Radiofrequency Treatments on Foot Functionality Index, Patient Satisfaction and Pain Scores in Plantar Fasciitis Patients
Brief Title: Effect of Radiofrequency Treatment in Plantar Fasciitis Patients
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Medical Doctor, Ankara University
Other Study IDs: 2024/202
Record Dates: First submitted 2024-05-18; First posted 2024-05-23 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2024-05

CONDITIONS: Fasciitis, Plantar
Keywords: Fasciitis, Plantar; Radiofrequency Therapy
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- posterior tibial nerve radiofrequency: posterior tibial nerve pulsed radiofrequency treatment
  Interventions: Procedure: posterior tibial nerve radiofrequency
- plantar fasciitis radiofrequency: calcaneal spur thermocoagulation radiofrequency treatment
  Interventions: Procedure: plantar fasciitis radiofrequency
- posterior tibial nerve and plantar fasciitis radiofrequency: posterior tibial nerve pulsed radiofrequency and calcaneal spur thermocoagulation radiofrequency treatment
  Interventions: Procedure: posterior tibial nerve radiofrequency; Procedure: plantar fasciitis radiofrequency

INTERVENTIONS:
Procedure: posterior tibial nerve radiofrequency — pulse radiofrequency at 45 V for 300 seconds at 42 degrees Celsius is applied to the posterior tibial nerve area. During the procedure, the temperature at the electrode tip is kept below 42°C. Following negative aspiration (in the absence of blood), 2 cc of 1% lidocaine + 4 mg dexamethasone is applied to the same area.
  Groups: posterior tibial nerve and plantar fasciitis radiofrequency; posterior tibial nerve radiofrequency
Procedure: plantar fasciitis radiofrequency — the spur area on the calcaneal bone is identified, and sensory and motor stimulations are applied using the RF cannula. If no sensory or motor response is elicited in the area, conventional radiofrequency at 45 V for 60 seconds at 80 degrees Celsius is applied to the spur area after confirming the placement of the RF cannula.
  Groups: plantar fasciitis radiofrequency; posterior tibial nerve and plantar fasciitis radiofrequency

SUMMARY:
In adults, chronic plantar fasciitis stands as the predominant cause of persistent heel discomfort.Usually, individuals depict a pulsating pain concentrated around the point of origin of the plantar fascia on the calcaneus. Numerous randomized and non-randomized studies have demonstrated the effectiveness of radiofrequency as a treatment modality for chronic plantar heel pain.In this study, our objective is to assess the impact of radiofrequency modalities applied to the posterior tibial nerve and/or the calcaneal spur area, guided by ultrasound, on patient satisfaction, pain scores, and functional improvement in individuals with chronic plantar fasciitis

DETAILED DESCRIPTION:
Chronic plantar fasciitis is the most common cause of chronic heel pain in adults. Typically, patients describe a throbbing pain localized around the origin of the plantar fascia on the calcaneus. This pain is often most severe when taking the first steps in the morning or rising after sitting. It typically improves with activity but worsens with prolonged activity. The primary aim of heel spur treatment is to alleviate pain and restore function. Surgical interventions are recommended for chronic plantar heel pain resistant to conservative options. However, surgery may be associated with prolonged recovery, and in one study, superiority over conservative treatment was not demonstrated. Radiofrequency has been shown to be an effective treatment method for chronic plantar heel pain in many randomized and non-randomized studies. In many studies, most of these procedures are applied blindly based on anatomical landmarks, with attention drawn in many studies to applications targeting the terminal branches of the posterior tibial nerve or the spur region. Only a few studies have been performed using fluoroscopy and ultrasound guidance. Ultrasound guidance offers several advantages over fluoroscopy and blind landmark techniques, especially in interventional procedures targeting neural and soft tissues. These advantages include the ability to visualize vascular and neural structures, very low risk of vascular-neural injury, absence of radiation exposure, and superiority in cases of anatomical variation. However, a common point in many studies related to plantar fasciitis is that applications are either directed to the spur area or to neural structures leading to the heel region. In this study, we aim to compare the effects of radiofrequency modalities applied to the posterior tibial nerve and/or calcaneal spur area under ultrasound guidance on patient satisfaction, pain scores, and patient functionality in cases of chronic plantar fasciitis (heel spur).

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old,
* Heel pain for at least 6 months and a diagnosis of plantar fasciitis confirmed by direct radiography and physical examination,
* Visual analog scale is 4 or more
* No response to conservative treatment (medical and physical medicine modalities)

Exclusion Criteria:

* History of trauma or calcaneus fracture,
* Osteoarthritis, Diabetes mellitus, chronic heart disease
* Presence of pregnancy,
* Pain due to peripheral neuropathy or ischemia
* Inability to tolerate injections in the heel area,
* Allergy to local anesthetics or steroids,
* Presence of an open wound on the side of the foot that the injection will be performed
* Local or systemic infection at the time of the procedure
* Previous steroid injection, radiofrequency application or ESWT (electroshock wave) treatment into the heel
* History of surgical intervention to the heel
* Presence of any functional limitation in the affected foot
* Presence of neurological, hepatic and/or metabolic diseases; dermatological infections, seronegative spondyloarthropathy, bleeding diathesis
* Failure to discontinue anticoagulant or antiaggregant within the specified periods
* Absence of follow-up throughout the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who are scheduled to receive radiofrequency tretament due to plantar fasciitis will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-07-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
pain severity | 1 and 3 months
  pain severity change by using Numeric Rating Scala will be observed before and at 1 week, 1, 3 months after the procedure.
  pain severity change by using Numeric Ratin Scala was observed 3 months after the procedure.The 11-point numerical scale ranges from '0', representing "no pain", to '10', representing extreme pain (e.g., "pain as bad as you can imagine" or "worst pain imaginable").
Patient satisfaction after the procedure | 1 and 3 months
  Patients will evaluate their satisfaction after the procedure as "satisfied", "uncertain" or "not satisfied".
functionallity | 1 and 3 months
  Functionality of foot will be observed at before the procedure and 1 week, 1, 3 months after the procedure. Foot functionalliy index will be used. Foot function index consists of 23 items with 3 subgroups: pain, disability and activity limitation. To calculate the subscales and total score, the scores of each item are summed, divided by the sum of the maximum scores of the items and multiplied by 100. Higher scores indicate more pain, disability, and activity limitation. The survey score varies between 0-100, and as the score increases, the disability increases.
medication use | 1 and 3 months
  number of medication use (nonsteroidal anttinflamatort drugs, opioids, muscle relaxants) wiil be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Hanzade A Unal, MD, Study Director — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Latt LD, Jaffe DE, Tang Y, Taljanovic MS. Evaluation and Treatment of Chronic Plantar Fasciitis. Foot Ankle Orthop. 2020 Feb 13;5(1):2473011419896763. doi: 10.1177/2473011419896763. eCollection 2020 Jan. PMID 35097359
- [Background] Li X, Zhang L, Gu S, Sun J, Qin Z, Yue J, Zhong Y, Ding N, Gao R. Comparative effectiveness of extracorporeal shock wave, ultrasound, low-level laser therapy, noninvasive interactive neurostimulation, and pulsed radiofrequency treatment for treating plantar fasciitis: A systematic review and network meta-analysis. Medicine (Baltimore). 2018 Oct;97(43):e12819. doi: 10.1097/MD.0000000000012819. PMID 30412072
- [Background] Wu YT, Chang CY, Chou YC, Yeh CC, Li TY, Chu HY, Chen LC. Ultrasound-Guided Pulsed Radiofrequency Stimulation of Posterior Tibial Nerve: A Potential Novel Intervention for Recalcitrant Plantar Fasciitis. Arch Phys Med Rehabil. 2017 May;98(5):964-970. doi: 10.1016/j.apmr.2017.01.016. Epub 2017 Feb 14. PMID 28209507
- [Background] Orhurhu V, Urits I, Orman S, Viswanath O, Abd-Elsayed A. A Systematic Review of Radiofrequency Treatment of the Ankle for the Management of Chronic Foot and Ankle Pain. Curr Pain Headache Rep. 2019 Jan 19;23(1):4. doi: 10.1007/s11916-019-0745-5. PMID 30661127